CLINICAL TRIAL: NCT00276419
Title: Topical Diclofenac for the Treatment of Noncyclic Breast Pain
Brief Title: Treatment of Breast Pain Using A Medication (Diclofenac) Applied to the Skin
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funds; FDA approved a topical form of diclofenac during study, no need to continue study of pharmacy-compounded drug.
Sponsor: Mayo Clinic (Other)
Responsible Party: Robin L. Smith, MD; principal investigator, Division of General Internal Medicine, Mayo Clinic, Rochester Minnesota
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 92-05
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Breast Pain; Non-cyclical Mastalgia; Surgical Scar-Related Breast Pain
MeSH Terms: conditions — Mastodynia | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo First, then Diclofenac (Arm A) (Experimental): Placebo for Diclofenac in topical cream applied to the skin three times daily for 10 weeks, then compounded topical Diclofenac cream applied to the skin three times daily for 10 weeks.
  Interventions: Drug: Diclofenac; Drug: Placebo
- Diclofenac First, then Placebo (Arm B) (Experimental): Compounded topical Diclofenac cream applied to the skin three times daily for 10 weeks, then placebo for Diclofenac in topical cream applied to the skin three times daily for 10 weeks.
  Interventions: Drug: Diclofenac; Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac — Compounded topical diclofenac cream applied to the skin three times daily for 10 weeks
  Other Names: Cambia; Cataflam; Voltaren; Voltarol; Zipsor
Drug: Placebo — Placebo for Diclofenac in topical cream applied to the skin three times daily for 10 weeks

SUMMARY:
The study was a randomized, double-blinded, crossover trial of topical diclofenac and placebo (10 weeks of each) for the treatment of noncyclic breast pain.

DETAILED DESCRIPTION:
A prospective, randomized, double-blinded crossover trial comparing topical diclofenac and placebo for 10 weeks in the treatment of 30 women with noncyclic mastalgia and surgical scar-related breast pain.

ELIGIBILITY:
Inclusion criteria

* Noncyclic mastalgia or surgical scar-related pain occurring at least 2 days per week and for which the patient desires treatment
* Duration of pain > 2 months (noncyclic mastalgia) or > 4 months (surgical scar-related pain)
* Age > 18 years
* Satisfactory breast examination and directed ultrasound at site of pain (all ages) within 12 months
* Satisfactory mammogram (all women > 30 years of age) within 12 months
* Negative pregnancy test (all women who are premenopausal and have not had hysterectomy or tubal ligation)

Exclusion criteria

* Cyclic mastalgia (as defined above)
* Duration of pain > 2 months (noncyclic mastalgia) or > 4 months (surgical scar-related pain)
* Abnormal breast examination or imaging (abnormality at the site of pain or for which biopsy or surgical consultation is recommended)
* Known pregnancy, lactation, positive pregnancy test, or anticipated pregnancy within 6 months
* Asthma, that has been aggravated by oral nonsteroidal antiinflammatory agents
* Allergy, to diclofenac or any nonsteroidal antiinflammatory agents
* Rash or open lesions at the site on the breast where the topical agent would be applied
* Incomplete or abnormal healing (surgical scar-related pain)
* History of gastrointestinal ulceration, renal dysfunction (creatinine > 1.5), hepatic disease (known liver disease or aspartate aminotransferase (AST) twice normal levels), congestive heart failure and uncontrolled hypertension (blood pressure > 140/90)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin L. Smith, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 Participants were recruited at the Mayo Clinic in Rochester Minnesota from June 2005 to May 2009. Seven subjects withdrew after randomization, prior to treatment, 6 in arm A, and 1 in arm B.
Period: First Intervention
Arm/Group | Placebo First, Then Diclofenac (Arm A) | Diclofenac First, Then Placebo (Arm B)
Started | 8 | 10
Completed | 7 | 8
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Wash-out Phase
Arm/Group | Placebo First, Then Diclofenac (Arm A) | Diclofenac First, Then Placebo (Arm B)
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Diclofenac (Arm A) | Diclofenac First, Then Placebo (Arm B)
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Diclofenac (Arm A) | Diclofenac First, Then Placebo (Arm B) | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Breast Pain
Description: Participants will complete a breast pain diary indicating the sensation of pain on a daily basis. The frequency of breast pain will be determined by the number of days per week that the subject recorded experiencing pain at 4 weeks and 10 weeks of each treatment.
Time Frame: 4 weeks, 10 weeks
Arm/Group | Placebo First, Then Diclofenac (Arm A) | Diclofenac First, Then Placebo (Arm B)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Severity of Breast Pain
Description: Severity will measured using a 100 mm visual analog scale (VAS). The VAS does not have any pre-set marks between the extremes. For the pain severity VAS, 0 means no pain and 100 means extreme pain. The investigator measures the written mark of the participant in mm, and records this for the value of pain severity. The severity of breast pain will be determined by the mean of breast pain scores (determined for all days and for days for which pain is greater than 0) at 4 weeks and 10 weeks of each treatment.
Time Frame: 4 weeks, 10 weeks
Arm/Group | Placebo First, Then Diclofenac (Arm A) | Diclofenac First, Then Placebo (Arm B)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Days of Pain During the 10 Week Treatment Periods
Description: Participants will complete a breast pain diary indicating the sensation of pain on a daily basis. Mean number of days with pain during each 10 week treatment period will be calculated.
Time Frame: Approximately 12 weeks and at 24 weeks after randomization
Arm/Group | Placebo First, Then Diclofenac (Arm A) | Diclofenac First, Then Placebo (Arm B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 22 weeks of the study.
Arm/Group | Placebo | Diclofenac
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Diclofenac (N=18)
Infection grade 2 (General disorders) | 1 (1) | 0 (0)
Dry skin of hand and scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of funds; the FDA approved a topical form of diclofenac during study, therefore there was no need to continue study of pharmacy-compounded drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No